CLINICAL TRIAL: NCT05840705
Title: Approach Modification for Total Knee Arthroplasty in Morbidly Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Saeed Younis, Lecturer of orthopaedics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54321askay
Record Dates: First submitted 2023-01-01; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Arthropathy; Incision, Surgical; Obesity, Morbid
Keywords: Total knee arthroplasty; obese
MeSH Terms: conditions — Joint Diseases; Surgical Wound; Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Total knee arthroplasty (Experimental)
  Interventions: Procedure: Small curved incision with apex lateral

INTERVENTIONS:
Procedure: Small curved incision with apex lateral — Small curved incision with apex lateral

SUMMARY:
The study provides a detailed description of a smaller incision with better visualization in total knee arthroplasty operations

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patients with body mass index more than 45 requiring total knee arthroplasty for any cause

Exclusion Criteria:

* candidates not meeting the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-08 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes | 3 years
  Knee society score
length of skin incision | 7 years
  lenght of skin incision in centimeters
operative time | 7 years
  Oprative time in minutes

SECONDARY OUTCOMES:
revision rate | 7 years
  no. of patients requiring revision
wound complications | 7 years
  Any reported wound complications
wound infection | 7 years
  No of patients with wound infection
Range of motion | 7 years
  Range of knee flexion and extension in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Saeed, Cairo, Egypt